CLINICAL TRIAL: NCT03334968
Title: Serum Prolidase Enzyme Activity as a Diagnostic Marker for Acute Ischemic Stroke
Brief Title: Prolidase Enzyme Activity in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Abdulkadir Tunc, Neurologist, Bezmialem Vakif University
Other Study IDs: StrokeProlidase
Record Dates: First submitted 2017-11-04; First posted 2017-11-07 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Stroke, Ischemic; Prolidase Deficiency
Keywords: Stroke; prolidase; prognosis; biomarker
MeSH Terms: conditions — Ischemic Stroke; Prolidase Deficiency; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Acute ischemic stroke patients
- Control group: Those served as control group

SUMMARY:
Stroke is a major cerebrovascular disease that causes significant burdens for human health and life, including high morbidity, mortality, and disability. Prolidase enzyme activity was found in various organs, such as the heart, brain, thymus, kidney, lung, pancreas, and spleen, and in plasma, leukocytes, erythrocytes, and dermal fibroblasts. An increase in collagen turnover is known to be correlated with increased prolidase enzyme activity. The aim of this study was to investigate whether SPA levels in AIS patients can be used as a potential diagnostic and prognostic marker. SPA levels were prospectively evaluated in 37 patients aged between 20 and 85 years who were admitted within 24 hours of the onset of AIS. The control group included 37 healthy volunteers of similar age without any disease.

DETAILED DESCRIPTION:
Ischemic stroke constitutes about 80-85% of all stroke cases and is caused by the interruption of cerebral blood flow due to a blood clot. Because of reactive oxygen species (ROS) production and its oxidative metabolite activity, the brain is highly sensitive to oxidative stress. This characteristic plays an important role in the pathogenesis of ischemic and hemorrhagic brain injuries .Prolidase, which is a cytosolic exopeptidase and a member of the matrix metalloproteinase (MMP) family, cleaves iminodipeptides from carboxy-terminal ends of proline or hydroxyproline and is actively involved in collagen metabolism. It has been shown that brain MMP activity is correlated with nutritive/oxidative stress and increases during reperfusion. Furthermore, in stroke patients, elevated serum MMP levels have been reported. Biomarkers that predict the outcome and occurrence of ischemic stroke are critically important for prevention and treatment .However, serum prolidase activity (SPA) has not been previously assessed in acute ischemic stroke (AIS) patients to our knowledge. Therefore, in this study, it's aimed to investigate whether SPA levels in AIS patients can be used as a potential diagnostic and prognostic marker.In the study, 37 patients aged between 20 and 85 years who were admitted within 24 hours of the onset of AIS were prospectively evaluated. The control group consisted of 37 healthy volunteers of similar age without any disease. A comprehensive physical examination was performed consisting of a neurological examination, blood biochemistry and blood count tests, electrocardiography, and a posterior-anterior chest X-ray for all patients. AIS patients underwent transthoracic echocardiography, multi-slice computed tomography (CT), and bilateral carotid-vertebral artery Doppler ultrasonography. National Institutes of Health Stroke Scale (NIHSS) scores, measured at 24 hours, 48 hours, and 28 days after stroke, were used to determine stroke severity.Ischemic stroke subtypes classification was done according to the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria, as cardioembolism, large-artery atherosclerosis, small artery occlusion, stroke of other determined cause, or undetermined cause. The measurement method for SPA was defined by Myara et al. The optimized method of Özcan et al. was used. Prolidase activity was evaluated with a spectrophotometric method, by measuring the proline levels. Briefly, 500 μL pre-incubation solution (50 mmol/L Tris hydrochloride buffer at power of hydrogen (pH) 7.8, with 1 mmol/L endogenous antioxidant glutathione (GSH), 5 mmol/L manganese(II) chloride (MnCl2), and 0.1% Triton X-100) and 100 μL serum were mixed; this mixture was then pre-incubated for 3 h at 37°C. A 100-μL volume of pre-incubation serum was added to 100 μL 144 mmol/L Gly-Pro solution, and this mixture was incubated for 30 min at 37°C. After the incubation, 1 ml 0.45 mol/L Trichloroacetic acid solution was added quickly to the incubation tube, and the incubation reaction was stopped. This mixture was centrifuged at 1500 rpm for 5 min, and 500 μL supernatant was removed.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 85
* admitted within 24 hours of the onset of acute ischemic stroke

Exclusion Criteria:

* patients with heart disease (such as myocardial infarction or heart failure
* chronic obstructive pulmonary disease,
* pulmonary embolism,
* pulmonary hypertension,
* tuberculosis,
* lung cancer,
* chronic renal failure,
* current hormone replacement treatment.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients WHO were evaluated in the tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Serum prolidase enzyme activity measurement | 24 hours
  Evaluation of serum prolidase enzyme activity in stroke patients and control group

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkadir TUNÇ, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gonullu H, Aslan M, Karadas S, Kati C, Duran L, Milanlioglu A, Aydin MN, Demir H. Serum prolidase enzyme activity and oxidative stress levels in patients with acute hemorrhagic stroke. Scand J Clin Lab Invest. 2014 Apr;74(3):199-205. doi: 10.3109/00365513.2013.873949. Epub 2014 Jan 23. PMID 24456419
- [Result] Verma AK, Raj J, Sharma V, Singh TB, Srivastava S, Srivastava R. Plasma Prolidase Activity and Oxidative Stress in Patients with Parkinson's Disease. Parkinsons Dis. 2015;2015:598028. doi: 10.1155/2015/598028. Epub 2015 Aug 9. PMID 26347150
- [Result] Tabur S, Oguz E, Eren MA, Korkmaz H, Savas E, Aksoy N, Sabuncu T. Serum prolidase activity is associated with non-diabetic metabolic syndrome. Diabetol Metab Syndr. 2014 Dec 17;6(1):142. doi: 10.1186/1758-5996-6-142. eCollection 2014. PMID 25540672
- [Result] Gasche Y, Copin JC, Sugawara T, Fujimura M, Chan PH. Matrix metalloproteinase inhibition prevents oxidative stress-associated blood-brain barrier disruption after transient focal cerebral ischemia. J Cereb Blood Flow Metab. 2001 Dec;21(12):1393-400. doi: 10.1097/00004647-200112000-00003. PMID 11740200
- [Result] Myara I, Charpentier C, Lemonnier A. Optimal conditions for prolidase assay by proline colorimetric determination: application to iminodipeptiduria. Clin Chim Acta. 1982 Oct 27;125(2):193-205. doi: 10.1016/0009-8981(82)90196-6. PMID 7139961
- [Result] CHINARD FP. Photometric estimation of proline and ornithine. J Biol Chem. 1952 Nov;199(1):91-5. No abstract available. PMID 12999819
- [Result] Danton GH, Dietrich WD. Inflammatory mechanisms after ischemia and stroke. J Neuropathol Exp Neurol. 2003 Feb;62(2):127-36. doi: 10.1093/jnen/62.2.127. PMID 12578222